CLINICAL TRIAL: NCT01231243
Title: Color Change and Sensitivity Level for In-office Bleaching With and Without a LED/Laser Device
Brief Title: Clinical Effectiveness of In-office Bleaching Activated With a LED/Laser Device
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Estadual de Ponta Grossa (Other)
Responsible Party: Principal Investigator, Alessandra Reis, PhD, Universidade Estadual de Ponta Grossa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ARAL001
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Tooth Discoloration
Keywords: tooth bleaching, bleaching agent, hydrogen peroxide
MeSH Terms: conditions — Tooth Discoloration | interventions — Tooth Bleaching; Hydrogen Peroxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 35% hydrogen peroxide control (Active Comparator): The tooth bleaching will be performed using a high hydrogen peroxide concentration (35%) without light-activation with LED/light device
  Interventions: Procedure: in-office bleaching with/without light
- 20% hydrogen peroxide (Active Comparator): The tooth bleaching will be performed with a low hydrogen peroxide concentration (20%) without light activation with a LED/laser device
  Interventions: Procedure: in-office bleaching with/without light
- 35% hydrogen peroxide + light (Experimental): The tooth bleaching will be performed with a high hydrogen peroxide concentration (35%) associated with LED/laser light activation
  Interventions: Procedure: in-office bleaching with/without light
- 20% hydrogen peroxide + light (Experimental): The tooth bleaching will be performed with a low hydrogen peroxide concentration (20%) associated with LED/laser light activation
  Interventions: Procedure: in-office bleaching with/without light

INTERVENTIONS:
Procedure: in-office bleaching with/without light — Two clinical sessions of tooth bleaching will be performed in each patient with a 1-week interval between them. In each session, three 15-min applications of the gel will be done using one of the two concentrations under investigation. In half of the sample of each concentration, the gel will be activated with a LED/laser device for a total of 3 min, as specified by the DMC manufacturer.
  Other Names: Tooth bleaching; Hydrogen peroxide; In-office bleaching; Light activation; Hydrogen peroxide concentration

SUMMARY:
There is a controversy in the dentistry literature about how the use of associated light to activate 35% hydrogen peroxide gel during in-office tooth bleaching may increase the bleaching effectiveness. The studies that demonstrated an increased level of bleaching using light activation employed lower hydrogen peroxide gels while the ones reporting no statistical difference employed higher hydrogen peroxide gels.

The hypothesis of this study is that the effectiveness of light activation tooth bleaching in dependent on the hydrogen peroxide concentration employed.

DETAILED DESCRIPTION:
The aim of this study is to compare the color change and tooth sensitivity of in-office bleaching using different hydrogen peroxide concentrations and with or without light activation. Sixty patients will be enrolled in this trial and divide equally into 4 groups according to the combination of the main factors hydrogen peroxide concentration (35% or 20%) or LED/laser activation (yes or no). Three 15-min applications will be performed in each clinical appointment. A LED/laser device will be used in the respective groups for three 1-min application with an interval of 2 min. The same procedure will be repeated one week later. The color change will be assessed after hte 1st and 2nd session, after 1 week and 6 months of the end of the treatment using a value-oriented shade Vita Classical and a spectrophotometer Easy Shade. The tooth sensitivity will be reported by patients using a 0 to 10 visual analog scale. The Student t test (α = .05) will be used to compare the tooth color changes and the intensity of tooth sensitivity between groups at baseline and immediately after the first and second bleaching appointments. The Fisher exact test and Student t test (α = .05), respectively, will be used to analyze the percentage of patients with tooth sensitivity and its intensity.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be at least 18 years old;
* Participants should have good general and oral health
* Participants should have six caries-free maxillary anterior teeth without restorations on the labial surfaces
* Participants should be willing to sign a consent form
* Participants should have central incisors darker than shade C2.

Exclusion Criteria:

* Participants that had undergone tooth-whitening procedures
* Participants that had labial anterior restorations, were pregnant or lactating.
* Participants with severe internal tooth discoloration (such as tetracycline stains, fluorosis, pulpless teeth).
* Participants with bruxism habits or any gross pathology in the mouth

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in color | at the 2-week recall
  The change in color will be measured using Vita Shade Classical scale at baseline and after the end of the bleaching protocol.
  A spectrophootometer Easy Shade will also be used and the coordinates of the CIELab system will be recorded.

SECONDARY OUTCOMES:
Prevalence and intensity of tooth sensitivity | 24-hours after the bleaching
  The visual analog scale will be used for patients to record their tooth sensitivity in a 0 to 10 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Reis, DDS, MS, Principal Investigator — Universidade Estadual de Ponta Grossa
Locations (1):
- School of Dentistry - Universidade Estadual de Ponta Grossa, Ponta Grossa, Paraná, Brazil